CLINICAL TRIAL: NCT00498355
Title: Effect of Ranibizumab on Refractory Macular Edema in Uveitis
Brief Title: Lucentis for Inflammatory Macular Edema Trial
Acronym: LIME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3872s
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Uveitis; Cytoid Macular Edema
Keywords: uveitis; cytoid macular edema; steroid; Lucentis
MeSH Terms: conditions — Uveitis | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental): 0.5 mg of ranibizumab by intravitreal injection at baseline and at monthly intervals for the following two months for a total of 3 injections. Afterwards, PRN injections for 9 months.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg of ranibizumab by intravitreal injection at baseline and at monthly intervals for the following two months for a total of 3 injections. Afterwards, PRN injections for 9 months.
  Other Names: Lucentis

SUMMARY:
Uveitis is an inflammation (swelling and irritation) inside the eye, affecting the uvea. The uvea is the layer of the eye between the sclera and the retina and provides most of the blood supply to the retina.

Uveitis is an important cause of visual loss. There are 30,000 new cases of legal blindness each year due to uveitis in the U.S. Sight-threatening complications associated with uveitis include macular edema, which may persist even when inflammation is controlled. The only current treatment for cystoid macular edema (CME) in uveitis patients is oral or regional steroid injections. For patients who don't respond to steroids or who are unable to tolerate steroid therapy, there are no other medical treatments.

The aim of this study is to determine if ranibizumab, an FDA-approved treatment for neovascular age-related macular degeneration, is an effective treatment for those patients with uveitis-induced CME who are unable to be treated with or non-responsive to steroids.

DETAILED DESCRIPTION:
Uveitis, an inflammation that affects the uvea (iris, ciliary body and choroid), is an important cause of visual loss. There are 30,000 new cases of legal blindness each year due to uveitis in the U.S. Sight-threatening complications associated with uveitis include macular edema, which may persist even when inflammation is controlled. The only current treatment for cystoid macular edema (CME) in uveitis patients is oral or regional steroid injections. For patients who don't respond to steroids or who are unable to tolerate steroid therapy, there are no other medical treatments.

The aim of the proposed research is to determine if ranibizumab is an effective treatment for those patients with uveitis-induced CME who are unable to be treated with or non-responsive to steroids. Ranibizumab is a recombinant, humanized monoclonal antibody antigen-binding fragment (Fab) that neutralizes all active forms of vascular endothelial growth factor (VEGF). VEGF is suspected to play a role in the loss of vascular integrity in the eye, which is thought to be involved in the pathogenesis of macular edema in the eyes of patients with uveitis. Ranibizumab was approved by the FDA for the treatment of neovascular age-related macular degeneration on June 30, 2006, and a number of published papers have shown efficacy for other causes of macular edema, including that due to diabetes mellitus.

The F. I. Proctor Foundation at UCSF will be enrolling 10 subjects 18 years of age or older with uveitis-induced CME to clinically evaluate the safety and effectiveness of ranibizumab administered monthly for three months followed by PRN monthly dosing (up to 12 months). The study will measure visual acuity, changes in foveal thickness on optical coherence tomography, and changes in cystoid macular edema by fluorescein angiography to determine the efficacy of ranibizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age ≥ 18 years
* A history of non-infectious uveitis with chronic cystoid macular edema (> 3 months duration)
* Foveal retinal thickness of ≥ 300 µM by OCT testing
* One prior trial of oral or regional steroid treatment for CME ≥ 30 days prior to study enrollment with persistent CME (≥ 300 µM foveal retinal thickness on OCT) or inability to use steroid injections due to a history of increased IOP above 30 mmHg thought to be due to topical steroid treatment or prior steroid injections
* Anterior chamber and vitreous inflammation at the trace or below level according to the standardized classification of inflammation
* BCVA at 4 m using the ETDRS chart of 20/40 to 20/400 (Snellen equivalent) in the study eye
* Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant, or premenopausal but not using adequate contraception
* Treatment for CME with oral or steroid injections, Macugen, or Avastin within 6 weeks prior to enrollment in this study. Study subjects will be allowed to continue their immunomodulatory treatment for uveitis throughout the study.
* Previous vitrectomy
* Active intraocular inflammation in the study eye (greater than trace anterior chamber or vitreous cells)
* Current vitreous hemorrhage
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Known allergy to any component of the study drug
* Intraocular pressure > 30 mm Hg despite treatment with glaucoma medications
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, the subject can become eligible.
* Major surgery planned during the next 6 months
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Unwilling or unable to follow or comply with all study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Acharya, MD MS, Principal Investigator — University of California, San Francisco
Locations (1):
- Proctor Foundation, UCSF, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the F.I. Proctor Foundation Uveitis Clinica at University of California San Francisco.
Groups:
- Ranibizumab for Macular Edema: This study was an open-label, single-center, prospective, nonrandomized interventional case series of 7 eyes in 7 patients with controlled uveitis and persistent visually significant macular edema.
Period: Overall Study
Arm/Group | Ranibizumab for Macular Edema
Started | 7
Completed | 6
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab for Macular Edema
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (15.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change at 3 Months in BSCVA From Baseline
Description: The outcome measure was mean best spectacle-corrected visual acuity (BSCVA). In this study, BSCVA was measured after trial frame manifest refraction, using high-contrast modified Bailey-Lovie (ETDRS) charts at 4 meters. The charts were placed in a retro-illuminated light box equipped with two 20-watt fluorescent tubes. The highest attainable 4-meter visual acuity score is 100 letters.
Time Frame: baseline and 3 months
Population: 6 patients completed all assessment points. One patient decided not to continue for nonmedical reasons, but they did complete the baseline, 1-week and 1-month assessment.
Measure: Mean (Full Range); unit: letters
Arm/Group | Ranibizumab for Macular Edema
Number analyzed (Participants) | 6
letters | 13 [3 to 24]

2. Secondary Outcome: The Median Change in Best Corrected Visual Acuity From 6 to12 Months
Time Frame: 6 to 12 months
Measure: Median (Full Range); unit: Letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 5
Letters | -2 [-6 to 2]

3. Secondary Outcome: The Mean Change in Foveal Retinal Thickness From Baseline at 7 Days, and at Months 3, 6, 9, and 12
Time Frame: 7 days, and at months 3, 6, 9, and 12
Measure: Mean (Full Range); unit: microns
Arm/Group | Ranibizumab
Number analyzed (Participants) | 7
microns
  Week 7 | -267 [-620 to -158]
  Month 3 | -356 [-1034 to -95]
  Month 6 | -354 [-1053 to -85]
  Month 9 | -243 [-941 to 222]
  Month 12 | -388 [-1026 to 12]

4. Secondary Outcome: The Incidence of Uveitis Flares (> 2+ Cells in the Anterior Chamber or Vitreous)
Time Frame: Study duration
Measure: Number; unit: uveitis flares
Arm/Group | Ranibizumab
Number analyzed (Participants) | 7
uveitis flares | 0

5. Secondary Outcome: The Incidence of Ocular and Non-ocular Adverse Events
Time Frame: Study duration
Measure: Number; unit: adverse events
Arm/Group | Ranibizumab
Number analyzed (Participants) | 7
adverse events | 4

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Ranibizumab for Macular Edema
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranibizumab for Macular Edema (N=7)
Subconjunctival Hemorrhage (Eye disorders) | 4 (4) — Transient subconjunctival hemorrhage, or burst blood vessel, after intravitreal injection.

LIMITATIONS AND CAVEATS:
Limitations of the study include a small sample size and lack of a control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No